CLINICAL TRIAL: NCT00970918
Title: Prevalence of Atherosclerotic Disease in Asian Subjects Not on Lipid-lowering Agents, But With at Least Two CVD Risk Factors
Brief Title: Study of Artery Conditions of 'At-risk' Asian People Not on Lipid-lowering Drugs
Acronym: CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Purpose: Screening
Other Study IDs: D3560L00092
Record Dates: First submitted 2009-08-25; First posted 2009-09-03 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Carotid Intima Media Thickness
MeSH Terms: conditions — Cardiovascular Diseases | interventions — C-Reactive Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Measurement of the Carotid Intima Media thickness; Biological: Blood sample testing for hs-CRP

INTERVENTIONS:
Procedure: Measurement of the Carotid Intima Media thickness — one time, radiological procedure on both sides of the neck
Biological: Blood sample testing for hs-CRP — one time, blood sample taking

SUMMARY:
The purpose of this study is to obtain the distribution of measurements of the intima media thickness of carotid arteries in people with high cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent.
* Patients with at least two CVD risk factors but not on lipid-lowering agents

Exclusion Criteria:

* Subjects with CHD, any conditions that may affect hs-CRP levels.
* Subjects on any lipid-lowering drug treatment within the last 3 months prior study entry.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2609 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Measurement of Carotid Intima Media Thickness of people with high risk of cardiovascular disease but not on lipid lowering drugs | IIMT measurements taken only once, either on Visit 1 or Visit 2 (time gap between V1 and V2 should be less than 3 months)

SECONDARY OUTCOMES:
Lipid profile of people with high risk of cardiovascular disease but not on lipid lowering drugs | Blood sampling only once, either on Visit 1 or Visit 2 (time gap between V1 and V2 should be less than 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Yeoman, MD, Study Director — Asia Pacific Regional Office, AstraZeneca Singapore Pte Ltd 8 Wilkie Road, #07-01 Wilkie Edge, Singapore 228095
Locations (19):
- China (2):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Shanghai, Shanghai Municipality
- India (3):
  - Research Site, Gūrgaon
  - Research Site, Jaipur
  - Research Site, Meerut
- Indonesia (4):
  - Research Site, Denpasar, Bali
  - Research Site, Bandung-Jawa, Barat
  - Research Site, Semarang-Jawa, Tengah
  - Research Site, Surabaya, Timur
- Research Site, Kuching, Sarawak, Malaysia
- Philippines (2):
  - Research Site, Manila, Manila
  - Research Site, Quezon City
- Research Site, Seoul, Seoul, South Korea
- Taiwan (3):
  - Research Site, Kaohsiung, Taipei
  - Research Site, Shilin, Taipei
  - Research Site, Taoyuan, Taipei
- Research Site, Patumwan, Bangkok, Thailand
- Vietnam (2):
  - Research Site, Hanoi, Hanoi
  - Research Site, Ho Chi Minh City, Ho Chi Min